CLINICAL TRIAL: NCT03747107
Title: Pharmacist and Data Driven Quality Improvement in Primary Care
Acronym: P-DQIP
Status: Completed | Type: Observational
Sponsor: University of Dundee (Other)
Collaborators: NHS Tayside (Other Government)
Responsible Party: Principal Investigator, Nicola Gray, Dr, University of Dundee
Other Study IDs: 2018PS02
Record Dates: First submitted 2018-11-12; First posted 2018-11-20 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Medication Safety
Keywords: primary care; prescribing safety; adverse drug event; drug therapy risk; pharmacist; general practice
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: P-DQIP — The 'intervention' is a health board quality improvement programme to be implemented across all practices in one Scottish NHS health board and comprises the following components: (i) Case finding via the P-DQIP informatics tool to identify patients with drug therapy risks for review; (ii) Decision support via the P-DQIP informatics tool to facilitate medication reviews; (iii) Practice pharmacists will be trained on the use of the P-DQIP informatics tool and instructed to target patients at risk of bleeding and hypoglycaemia first (iv) Ongoing performance feedback. Practices and locality pharmacists will be able to access reports on review activity and targeted prescribing; (v) promotion of the P-DQIP tool and intervention among GP practices. The P-DQIP intervention will be evaluated in all NHS Tayside practices who agree to share their data for monitoring and evaluation purposes.

SUMMARY:
P-DQIP is an intervention to improve prescribing safety in primary care. The 'intervention' is a health board quality improvement programme that will be implemented across all practices in one National Health Service (NHS) board in Scotland (Tayside), and comprises the following components:

i. Case finding of patients with drug therapy risks via the P-DQIP informatics tool ii. Decision support for clinicians when conducting medication reviews via the P-DQIP informatics tool iii. Support from practice pharmacists in reviewing and managing targeted patients iv. Ongoing performance feedback via the P-DQIP informatics tool v. Promotion of the P-DQIP tool and intervention among general practices. The P-DQIP intervention will be evaluated in all NHS Tayside practices who agree to share their data for monitoring and evaluation purposes.

DETAILED DESCRIPTION:
P-DQIP is an intervention to improve prescribing safety in primary care. The 'intervention' is a health board quality improvement programme that will be implemented across all practices in NHS Tayside. The study is therefore a service evaluation of an NHS Tayside-led initiative, which comprises the following components:

i. Case finding. The P-DQIP informatics tool will be added to medicines management software (the Scottish Therapeutics Utility), which is already installed in all general practices in NHS Scotland. The P-DQIP tool can be accessed by General Practitioners (GPs) and other clinicians in the practice including Health Board employed primary care pharmacists 'attached' to practices. The core of the tool is a set of indicators of high-risk prescribing to identify patients at high risk of drug related harm. The indicators have been developed by The Scottish Government's Polypharmacy working group.

ii. Decision support. The P-DQIP tool provides structured information on patients' medical and medication histories and highlights specific drug therapy risks for consideration by the reviewing clinician. All decision making remains at the discretion of the reviewing clinician.

iii. Pharmacist support. Teams of practice pharmacists working in practices within the same locality will be invited to participate in a half-day workshop, in which they will be trained on the use of the P-DQIP informatics tool. A total of 8 to 12 workshops will be conducted. The workshop will be facilitated by the P-DQIP project team. As part of the workshop, locality pharmacist teams will be encouraged to plan the P-DQIP work and to agree targets. They will be instructed to introduce the P-DQIP pogramme in a stepwise fashion, targeting patients at risk of bleeding and hypoglycaemia first.

iv. Ongoing performance feedback. Practices and locality pharmacists will be able to access reports on the number of reviews conducted and the numbers of patients with targeted high-risk prescribing via the P-DQIP informatics tool.

v. Promotion of the P-DQIP tool and intervention among GP practices. GP clusters will be offered a visit by the lead pharmacist for the programme, who will provide background and rationale for the P-DQIP programme, demonstrate the functionalities of the P-DQIP informatics tool and encourage collaboration in reviewing and managing targeted drug therapy risks with pharmacists.

ELIGIBILITY:
Inclusion Criteria:

* General practices in NHS Tayside, who use the Vision electronic medical record software and agree to the extraction of data from medical records for monitoring and evaluation purposes

Exclusion Criteria:

* General practices using electronic medical record software other than Vision

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All general practices in NHS Tayside, who use the Vision electronic medical record software and agree to the extraction of data from medical records for monitoring and evaluation purposes
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Initially targeted drug therapy risks in patients aged 75 years or older | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  Denominator definition: No. of patients aged 75 years or older meeting one or more denominator definitions as specified under 'Other Pre-specified Outcomes' P001 to P011; Numerator definition: No. of denominator patients meeting one or more numerator definitions as specified under 'Other Pre-specified Outcomes' P001 to P011

SECONDARY OUTCOMES:
All targeted drug therapy risks in patients aged 75 years or older (patient count) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  Denominator definition: No. of patients aged 75 years or older meeting one or more denominator definitions as specified under 'Other Pre-specified Outcomes' P001 to P046; Numerator definition: No. of denominator patients meeting one or more numerator definitions as specified under 'Other Pre-specified Outcomes' P001 to P046
All targeted drug therapy risks in patients aged 75 years or older (indicator count) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  Denominator definition: No. of patients aged 75 years or older meeting one or more denominator definitions as specified under 'Other Pre-specified Outcomes' P001 to P046; Numerator definition: No. of indicators specified under 'Other Pre-specified Outcomes' P001 to P046 triggered by denominator patients
Initially targeted drug therapy risks in younger patients | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  Denominator definition: No. of patients aged <75 years meeting one or more denominator definitions as specified under 'Other Pre-specified Outcomes' P001 to P011; Numerator definition: No. of denominator patients meeting one or more numerator definitions as specified under 'Other Pre-specified Outcomes' P001 to P011;
All targeted drug therapy risks in younger patients (patient count) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  Denominator definition: No. of patients aged <75 years meeting one or more denominator definitions as specified under 'Other Pre-specified Outcomes' P001 to P046; Numerator definition: No. of denominator patients meeting one or more numerator definitions as specified under 'Other Pre-specified Outcomes' P001 to P046
All targeted drug therapy risks in younger patients (indicator count) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  Denominator definition: No. of patients aged <75 years meeting one or more denominator definitions as specified under 'Other Pre-specified Outcomes' P001 to P046; Numerator definition: No. of indicators specified under 'Other Pre-specified Outcomes' P001 to P046 triggered by denominator patients
'Ongoing' versus 'new' drug therapy risks ('Ongoing') | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  Denominator definition: No. of patients aged 75 years or older meeting one or more denominator definitions specified under 'Other Pre-specified Outcomes' P001 to P011, who have met one or more numerator definitions specified under 'Other Pre-specified Outcomes' P001 to P011 in the previous 57 to 364 days; Numerator definition (Old): No. of denominator patients meeting one or more numerator definitions specified under 'Other Pre-specified Outcomes' P001 to P011
'Ongoing' versus 'new' drug therapy risks ('New') | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  Denominator definition: No. of patients aged 75 years or older meeting one or more denominator definitions specified under 'Other Pre-specified Outcomes' P001 to P011, who have NOT met any numerator definitions specified under 'Other Pre-specified Outcomes' P001 to P011 in the previous 57 to 364 days; Numerator definition: No. of denominator patients meeting one or more numerator definitions specified under 'Other Pre-specified Outcomes' P001 to P011
Electrolyte disturbances | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  Denominator definition: No. of patients aged <75 years meeting one or more denominator definitions as specified under 'Other Pre-specified Outcomes' P047 to P050; Numerator definition: No. of indicators specified under 'Other Pre-specified Outcomes' P047 to P050 triggered by denominator patients
Related unscheduled care events (1) - Bleeding | Measured at intervals of 12 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  Denominator definition: No. of patients aged 75 years or older; Numerator definition: No. of denominator patients who had an unscheduled care event with bleeding in the previous 84 days
Related unscheduled care events (2) - Hypoglycaemia, falls, fractures | Measured at intervals of 12 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  Denominator definition: No. of patients aged 75 years or older; Numerator definition: No. of denominator patients who had an unscheduled care event with hypoglycaemia, a fall or a fracture in the previous 84 days
Related unscheduled care events (3) - Any potentially drug related events | Measured at intervals of 12 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  Denominator definition: No. of patients aged 75 years or older; Numerator definition: No. of denominator patients who had an unscheduled care event in the previous 84 days with any of the following: Hypoglycaemia, fall, fracture, bleeding, heart failure, bradycardia, acute kidney injury, constipation, dehydration, hyperkalaemia, hyponatraemia, urinary retention, delirium) in the previous 84 days
Unrelated unscheduled care events | Measured at intervals of 12 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  Denominator definition: No. of patients aged 75 years or older; Numerator definition: No. of denominator patients who had an unscheduled care event in the previous 84 days with an unrelated ambulatory care sensitive admission (Appendicitis, pancreatitis, cholecystitis, cancer, cellulitis)

OTHER OUTCOMES:
Individual indicators (P001) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  P001 - Denominator definition: No. of patients aged 75 and older; Numerator definition: No. of denominator patients with any non-topical non-steroidal anti-inflammatory drug (NSAID) issued in last 56d and NO gastro-protection issued in last 84d
Individual indicators (P002) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  P002 - Denominator definition: No. of patients aged 65 to 74 and gastrointestinal ulcer or issued an antiplatelet, oral anticoagulant or oral corticosteroid in last 56d; Numerator definition: No. of denominator patients with any non-topical NSAID issued in last 56d and NO gastro-protection issued in last 84d
Individual indicators (P003) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  P003 - Denominator definition: No. of patients aged 65 or older and aspirin issued in last 84d; Numerator definition: No. of denominator patients with clopidogrel issued in last 56d and NO gastro-protection issued in last 84d
Individual indicators (P004) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  P004 - Denominator definition: No. of patients with previous gastrointestinal ulcer; Numerator definition: No. of denominator patients with antiplatelet issued in last 56d and NO gastro-protection issued in last 84d
Individual indicators (P005) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  P005 - Denominator definition: No. of patients with an oral anticoagulant issued in last 84d; Numerator definition: No. of denominator patients with an antiplatelet issued in last 56d and NO gastro-protection issued in last 84d
Individual indicators (P006) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  P006 - Denominator definition: No. of patients with any of the following: Chronic kidney disease (CKD) stage 4 or 5 or latest estimated glomerular filtration rate (eGFR)<30ml/min (in previous 364 days); Numerator definition: No. of denominator patients with direct thrombin inhibitor issued in last 56d
Individual indicators (P007) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  P007 - Denominator: One of the following: CKD stage 5 or latest eGFR showing eGFR<15ml/min (in previous 364d); Numerator: Factor Xa inhibitor issued in last 56d
Individual indicators (P008) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  P008 - Denominator definition: No. of patients with an oral anticoagulant issued in last 84d; Numerator definition: No. of denominator patients with latest SBP>160 or latest DBP>100 BP (in previous 364 days)
Individual indicators (P009) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  P009 - Denominator definition: No. of patients with insulin issued in last 84d; Numerator definition: No. of denominator patients with no glucose test strips issued in last 56d
Individual indicators (P010) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  P010 - Denominator definition: No. of patients with diabetes type 2 and aged 75 or older or dementia; Numerator definition: No. of denominator patients with insulin or an oral hypoglycaemic drug other than metformin issued in last 56d and last glycated haemoglobin (HbA1c)<53 (7.0%) (in previous 364d)
Individual indicators (P011) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  P011 - Denominator definition: No. of patients Diabetes type 2 and aged 65 to 74 without dementia; Numerator definition: No. of denominator patients with insulin or an oral hypoglycaemic drug other than metformin issued in last 56d and last HbA1c<48 (6.5%) (in previous 364d)
Individual indicators (P012) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  P012- Denominator definition: No. of patients with an oral nitrate or nicorandil issued in last 84d; Numerator definition: No. of denominator patients with phosphodiesterase type-5 inhibitor issued in last 56d
Individual indicators (P013) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  P013- Denominator definition: No. of patients with heart failure; Numerator definition: No. of denominator patients with a glitazone issued in last 56d
Individual indicators (P014) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  P014- Denominator definition: No. of patients heart failure; Numerator definition: No. of denominator patients with any non-topical NSAID issued in last 56d
Individual indicators (P015) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  P015- Denominator definition: No. of patients with heart failure or issued a beta blocker in the previous 84d; Numerator definition: No. of denominator patients with verapamil or diltiazem issued in last 56d
Individual indicators (P016) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  P016- Denominator definition: No. of patients with heart failure without atrial fibrillation, CKD stage ≥3, latest eGFR<60ml/min (in previous 365 days) or verapamil issued in last 84d; Numerator definition: No. of denominator patients with digoxin tablets >125mcg strength issued in last 56d
Individual indicators (P017) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  P017- Denominator definition: No. of patients with beta blocker, acetylcholine esterase inhibitor or digoxin issued in last 84d; Numerator definition: No. of denominator patients with last pulse <60bpm
Individual indicators (P018) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  P018- Denominator definition: No. of patients with CKD stage 5 or latest eGFR<10ml/min (in previous 365d); Numerator definition: No. of denominator patients with colchicine issued in last 56d
Individual indicators (P019) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  P019- Denominator definition: No. of patients with methotrexate issued in last 84d; Numerator definition: No. of denominator patients with methotrexate 2.5mg strength issued and methotrexate 10mg strength issued in last 56d
Individual indicators (P020) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  P020- Denominator definition: No. of patients with methotrexate issued in last 84d; Numerator definition: No. of denominator patients with trimethoprim issued in last 56d and trimethoprim issued in last 57 to 112 days
Individual indicators (P021) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  P021- Denominator definition: No. of patients with one or more of the following risk factors for Acute Kidney Injury (AKI):
  * diuretic issued in last 84d and ACEI or ARB issued in last 84d
  * CKD stage 4 or 5 or latest eGFR<30ml/min (in previous 364d)
  * ACEI or ARB issued in last 84d and CKD stage 3 or latest eGFR 30 to 59ml/min (in previous 364d) in last 84d
  * diuretic issued in last 84d and CKD stage 3 or latest eGFR 30 to 59ml/min (in previous 364d) in last 84d; Numerator definition: No. of denominator patients with Any non-topical NSAID issued in last 56d
Individual indicators (P022) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  P022- Denominator definition: No. of patients with CKD stage 4 or 5 or latest eGFR <30 ml/min (in previous 365 days) or ACEI or ARB issued in last 84d; Numerator definition: No. of denominator patients with potassium salt issued in last 56d
Individual indicators (P023) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  P023- Denominator definition: No. of patients with angiotensin converting enzyme inhibitor (ACEI) or angiotensin receptor blocker (ARB) issued in last 84d; Numerator definition: No. of denominator patients with ACEI and ARB issued in previous 56d
Individual indicators (P024) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  P024- Denominator definition: No. of patients with ACEI or ARB issued in last 84d and no history of CKD stage 4 or 5 and latest eGFR >=30 ml/min or unknown (in previous 364d); Numerator definition: No. of denominator patients with potassium sparing diuretic and aliskiren issued in last 56d
Individual indicators (P025) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  P025- Denominator definition: No. of patients CKD stage 4 or 5 or latest eGFR <30 ml/min (in previous 364d); Numerator definition: No. of denominator patients with potassium sparing diuretic or aliskiren issued in last 56d
Individual indicators (P026) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  P026- Denominator definition: No. of patients with CKD stage 4 or 5 or latest eGFR <30 ml/min (in previous 364d); Numerator definition: No. of denominator patients with trimethoprim issued in last 56d
Individual indicators (P027) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  P027- Denominator definition: No. of patients with digoxin issued in the last 84d; Numerator definition: No. of denominator patients with latest potassium <3.0 mmol/L (in previous 364 d)
Individual indicators (P028) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  P028- Denominator definition: No. of patients with CKD stage 4 or 5 or latest eGFR <30 ml/min (in previous 364d); Numerator definition: No. of denominator patients with metformin issued in last 84d
Individual indicators (P029) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  P029- Denominator definition: No. of patients Aged 75 or older without heart failure; Numerator definition: No. of denominator patients with last systolic blood pressure (SBP) <110 and last diastolic blood pressure (DBP)<65 and any of the following issued in last 56d: ACEI, ARB, beta blocker, thiazide, calcium channel blocker, alpha blocker, oral nitrate, centrally acting antihypertensive drug
Individual indicators (P030) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  P030- Denominator definition: No. of patients with dementia and hypertension; Numerator definition: No. of denominator patients with Last SBP <130 and last DBP<75 and two or more of the following issued in last 56d: ACEI, ARB, beta blocker, thiazide, calcium channel blocker, alpha blocker, oral nitrate, centrally acting antihypertensive drug
Individual indicators (P031) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  P031- Denominator definition: No. of patients aged 65 years or older with dementia; Numerator definition: No. of denominator patients with antipsychotic issued in last 56d
Individual indicators (P032) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  P032- Denominator definition: No. of patients who are female and have previous venous thromboembolism; Numerator definition: No. of denominator patients with Oestrogen issued in last 56d
Individual indicators (P033) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  P033- Denominator definition: No. of patients with atrial fibrillation (AF) and C(ardiac failure)H(ypertension)A(ge)D(iabetes)S(troke/TIA)VASc(ular disease history) score >=3; Numerator definition: No. of denominator patients with NO oral anticoagulant issued in last 56d
Individual indicators (P034) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  P034- Denominator definition: No. of patients with asthma without chronic obstructive pulmonary disease (COPD) and a short acting beta agonist (SABA) issued in last 84d; Numerator definition: No. of denominator patients with non-cardio-selective beta blocker issued in last 56d
Individual indicators (P035) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  P035- Denominator definition: No. of patients aged 75 years and older and an oral steroid issued in last 84d and in the last 85 to 168 days; Numerator definition: No. of denominator patients with no bisphosphate, vitamin D or calcium issued in last 56d
Individual indicators (P036) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  P036- Denominator definition: No. of patients with dementia; Numerator definition: No. of denominator patients with two or more drugs with significant sedating or anticholinergic effects issued in previous 56d (excluding drugs only used for epilepsy)
Individual indicators (P037) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  P037- Denominator definition: No. of patients with no dementia and aged 65 to 74 years; Numerator definition: No. of denominator patients with THREE or more drugs with significant sedating or anticholinergic effects issued in previous 56d (excluding drugs only used for epilepsy)
Individual indicators (P038) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  P038- Denominator definition: No. of patients with no dementia and aged 75 years or older; Numerator definition: No. of denominator patients with two or more drugs with significant sedating or anticholinergic effects (excluding drugs only used for epilepsy)
Individual indicators (P039) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  P039- Denominator definition: No. of patients with opioid issued in last 84d; Numerator definition: No. of denominator patients issued an opioid in last 56d and issued opioids at an average daily dose equivalent to >180mg morphine per day over the previous 182d
Individual indicators (P040) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  P040- Denominator definition: No. of patients with gabapentin or pregabalin issued in last 84d; Numerator definition: No. of denominator patients issued gabapentin or pregabalin in the last 56d and issued gabapentin or pregabalin at an average daily dose of >4800mg gabapentin per day over the previous 182d
Individual indicators (P041) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  P041- Denominator definition: No. of patients with lithium issued in last 84d; Numerator definition: No. of denominator patients with an NSAID issued in the last 56d
Individual indicators (P042) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  P042- Denominator definition: No. of patients with lithium issued in last 84d; Numerator definition: No. of denominator patients with thiazide diuretic issued in previous 56d and no thiazide diuretic issued in previous 57 to 112 days
Individual indicators (P043) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  P043- Denominator definition: No. of patients with levodopa issued in last 84d; Numerator definition: No. of denominator patients with prochlorperazine issued in last 56d and previous 57 to 112d or metoclopramide issued in last 56d and previous 57 to 112d
Individual indicators (P044) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  P044- Denominator definition: No. of patients aged 65 years or older; Numerator definition: No. of denominator patients with metoclopramide issued in last 56 and in the previous 57 to 112d
Individual indicators (P045) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  P045- Denominator definition: No. of patients with a history of breast cancer; Numerator definition: No. of denominator patients with oestrogen issued in last 56d
Individual indicators (P046) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  P046- Denominator definition: No. of female patients aged 60 years or older; Numerator definition: No. of denominator patients with estrogen issued in last 56d
Individual indicators (P047) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  P047- Denominator definition: No. of patients with thiazide or a loop diuretic issued in the last 84d; Numerator definition: No. of denominator patients with latest potassium <3.0 mmol/L (in previous 364 d)
Individual indicators (P048) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  P048- Denominator definition: No. of patients with selective serotonin reuptake inhibitor (SSRI), thiazide or loop diuretic issued in last 84d; Numerator definition: No. of denominator patients with latest sodium <130 mmol/l (in previous 364 days)
Individual indicators (P049) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  P049- Denominator definition: No. of patients with a thiazide issued in last 84d; Numerator definition: No. of denominator patients with latest calcium >2.65 mmol/L (in previous 364 days)
Individual indicators (P050) | Measured at intervals of 8 weeks over a period of 18 months prior to and subsequent to the start date. The measurement on the start date will be excluded from analyses to account for the availability of a test version of the P-DQIP tool since Sept 2018
  P050- Denominator definition: No. of patients with ACEI or ARB, potassium sparing diuretic, aldosterone antagonist, aliskiren or potassium supplement issued in previous 84d; Numerator definition: No. of denominator patients with latest potassium >5.5mmol/L (in previous 364 days)

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Dreischulte, Principal Investigator — University of Dundee/NHS Tayside
Locations (1):
- NHS Tayside, Dundee, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No
We cannot agree to sharing individual participant data, since we do not own the data.